CLINICAL TRIAL: NCT02944058
Title: Plate Fixation Versus Intramedullary Nailing of 3 and 4 Part Proximal Humerus Fractures. A RCT
Brief Title: Plate Fixation Versus Intramedullary Nailing of 3 and 4 Part Proximal Humerus Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Asbjorn Aroen, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/626
Record Dates: First submitted 2016-10-17; First posted 2016-10-25 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Shoulder Fractures; Humeral Fractures, Proximal
Keywords: Multiloc; Philos; Locking plate; Straight nail; Randomized controlled trial; 3 and 4 part fractures
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Philos plate (Active Comparator): Intervention is surgery with Philos plate
  Interventions: Procedure: Philos plate
- Multiloc nail (Active Comparator): Intervention is surgery with Multiloc nail
  Interventions: Procedure: Multiloc nail

INTERVENTIONS:
Procedure: Multiloc nail — Intervention is surgery with Multiloc nail
  Arms: Multiloc nail
Procedure: Philos plate — Intervention is surgery with Philos plate
  Arms: Philos plate

SUMMARY:
The purpose of the project is to compare the management of 3 and 4 part proximal humerus fractures (PHF) with an angular stable plate (Philos) with that of an intramedullary nail (Multiloc) in light of complications, radiological, economical, functional and clinical outcome.

DETAILED DESCRIPTION:
Randomized controlled trial (RCT) from Akershus University Hospital in Norway. Randomization between two implants. The investigators will use deltopectoral or deltoid split as surgical access. All patients will have calcar screws and cuff sutures. When lack of bone for example after decompressing valgus compressed fractures, a bone-substitute might be used in the surgeons preference. Follow up in outpatient clinic at 6, 12, 52 and 104 weeks, but also a 5 year follow up is planned. Postoperative radiographs of both shoulders and CT of operated shoulder will be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years
2. Severe displacement, defined as malposition of at least 45⁰ of angular deviation in valgus or 30⁰ in varus in true frontal projection, regardless of whether the fracture is impacted or not. Fractures with more than 50% displacement of the head against the surgical neck
3. The greater or lesser tubercles must be fractured in a 3 or 4-part fracture. The degree of displacement is not critical for inclusion.

Exclusion Criteria:

Exclusion criteria:

1. Fracture more than 3 weeks' old
2. Caput humeri just a thin shell or split
3. Ipsilateral damage that will influence the recovery and scoring systems
4. Incapability to protect osteosynthesis, i.e. use of crutches because of injury to lower extremity.
5. Pathological fracture
6. Neurovascular injury
7. Open fracture
8. Noncompliance
9. Congenital anomaly
10. Ongoing infectious process around the incision site for plate osteosynthesis
11. Systemic disease that may influence healing processes or scoring systems (RA/MS)
12. Fracture dislocation
13. Substance abuse
14. Inability to read and understand Norwegian
15. Patients not residing in our catchment area
16. Patients with too small humerus diameter to use a nail
17. Patient not able to commit and understand written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2023-10-24 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand (DASH) Score (questionnaire) Disability of the arm, shoulder and arm score (DASH score) | 5 years
  Quick Dash (questionnaire) the first 6 weeks after surgery, then DASH score (questionnaire for patients to fill out) in follow ups

SECONDARY OUTCOMES:
Constant score (questionnaire) | 5years
  A questionnaire for the doctor or the physiotherapist to fill out, including registration of: Pain, Power, Range of motion and ADL (x/100, where 100 is best score)
Radiological complications | 5 years
  Plate cutout, Nail migration, screw cutout, Reduction of Head shaft angle (HSA)/ Varus subsidence,
Complications | 5 years
  Infection, Avascular necrosis, thrombosis, nerve compression or damage, Pseudoarthrosis
Health economy | 5 years
  Registration of visits to doctor, physiotherapist, sick leave, re-operations

CONTACTS AND LOCATIONS:
Overall Officials: Asbjorn AAroen, PhD MD, Study Director — Akershus University Hospital, orthopedic unit
Locations (1):
- Akershus University hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available within 6 months of study completion

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196